CLINICAL TRIAL: NCT01680887
Title: A Phase II, Randomized, Double-Blind Trial of Varenicline for the Treatment of Cocaine Dependence
Brief Title: A Phase II Trial of Varenicline for the Treatment of Cocaine Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 814643
Record Dates: First submitted 2012-08-28; First posted 2012-09-07 (Estimated); Results first posted 2019-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-07

CONDITIONS: Cocaine Dependence
Keywords: Cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varenicline (Experimental): Oral 1.0 mg BID.
  Interventions: Drug: Varenicline
- Placebo (Placebo Comparator): Oral 1.0 mg BID.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline
  Other Names: Chantix
  Arms: Varenicline
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a double-blind placebo-controlled clinical trial (n = 156) of varenicline for the treatment of cocaine dependence that utilizes contingency management to promote treatment attendance.

DETAILED DESCRIPTION:
Background: Varenicline is a medication approved for the treatment of Tobacco Use Disorder. It is a partial agonist at α2β4 nicotinic acetyl choline receptors and a full agonist at α7 nicotinic acetyl choline receptors. By its effects on cholinergic activity at α7 and α2β4 receptors, varenicline may reduce dopaminergic and glutamatergic activity in the midbrain, and reduce symptoms of Cocaine Use Disorder. A preliminary trial of varenicline in human cocaine users suggested that varenicline treatment was associated with reductions in cocaine use. The current trial was intended to confirm these promising preliminary results.

Methods: This was a 12-week, double blind, placebo controlled parallel group clinical trial involving 156 DSM IV cocaine dependent subjects. Subjects received 2 mg of varenicline or identical placebo each day along with weekly individual cognitive behavioral relapse prevention psychotherapy. The primary outcome measure was cocaine use measured by by thrice weekly urine drug screens. Additional outcome measures included cocaine withdrawal symptoms measured by the Cocaine Selective Severity Assessment (CSSA) End of study cocaine abstinence was analyzed using a Chi-square test.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, 18 to 65 years old.
2. Meets DSM-IV criteria for Cocaine Dependence, as determined by the Structured Clinical Interview for DSM-IV (SCID).
3. Live within a commutable distance of the Treatment Research Center (TRC) at the Penn/VA Center for Studies of Addiction, University of Pennsylvania. We define this to be a distance within the service area of Septa, within an hour drive, or a distance that both the patient and Principal Investigator (PI) find acceptable.
4. Understands and signs the informed consent.

Exclusion Criteria:

1. Current DSM-IV diagnosis of any psychoactive substance dependence other than cocaine, alcohol, or nicotine dependence, as determined by the SCID.
2. Subject is, in the investigator's opinion, at risk of requiring medical detoxification for alcohol dependence during the study.
3. Concomitant treatment with psychotropic medications.
4. Current gambling problems. This will be assessed by the patient's self-report.
5. Patients mandated to treatment based upon a legal decision or as a condition of employment who will use participation in this study to fulfill to their court mandated treatment requirement.This will be assessed by the patient's self-report.
6. Current severe psychiatric symptoms, e.g., psychosis, dementia, suicidal or homicidal ideation, mania or depression requiring antidepressant therapy in the opinion of the Principal Investigator (PI).
7. Use of any investigational medication within the past 30 days.
8. Subject has serious heart, lung, kidney, immune system, GI tract (ulcerative colitis, regional enteritis, or gastrointestinal bleeding) disease.
9. Current use of naltrexone, disulfiram, modafinil, stimulants, haloperidol, benzodiazepines or anticonvulsants.
10. Known hypersensitivity to varenicline.
11. Patients with known AIDS or other serious illnesses that may require hospitalization during the study.
12. Female subjects who are pregnant or lactating, or female subjects of child-bearing potential who are not using acceptable methods of birth control. Acceptable methods of birth control include:

    1. barrier (diaphragm or condom) with spermicide
    2. intrauterine progesterone contraceptive system
    3. levonorgestrel implant
    4. medroxyprogesterone acetate contraceptive injection
    5. oral contraceptives
    6. tubal ligation.
13. Patients with impaired renal function as indicated by corrected creatinine clearance below 60 ml/min as determined by the modified Cockcroft equation (CDC, 1986).
14. Clinical laboratory tests (CBC, blood chemistries, urinalysis) outside normal limits that are clinically unacceptable to the Medical Director. EKG 1st degree heart block, sinus tachycardia, left axis deviation, and nonspecific ST or T wave changes are allowed; liver function tests [LFTs] <5 x ULN are acceptable).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2012-08; Primary Completion 2018-01 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle M Kampman, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Treatment Research Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of Pennsylvania Center for Studies of Addictions — http://www.med.upenn.edu/csa/

RESULTS

PARTICIPANT FLOW:
Groups:
- Varenicline: Oral 1.0 mg BID.
  Varenicline
- Placebo: Oral 1.0 mg BID.
  Placebo
Period: Overall Study
Arm/Group | Varenicline | Placebo
Started | 80 | 76
Completed | 51 | 52
Not Completed | 29 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 80 | 76 | 156
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 80 | 75 | 155
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 34
  Male | 62 | 60 | 122
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 68 | 68 | 136
  White | 12 | 8 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 80 | 76 | 156

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Report no Cocaine Use and Have no Cocaine Positive Urine Drug Screens in the Chantix Group Versus the Placebo Group Comparator During the Last Three Weeks of the Trial
Description: Number of subjects with cocaine abstinence as measured through three-times-weekly urine benzoylecgonine (BE) levels in urine drug screen (UDS) and self-reports of use from the Time Line Follow Back. UDS results and TLFB reports combined to yield weekly use/no-use indicators for each week of treatment.
Time Frame: weeks 11,12,13 of the trial
Population: all subject
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 80 | 76
Participants | 6 | 7
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Test type: Superiority; p = .403, Chi-squared

2. Secondary Outcome: Average Weekly Cocaine Craving Scores Varenicline Group Versus the Placebo Group Comparator
Description: As measured by average weekly scores for cocaine craving on the brief substance craving scale combining cocaine craving frequency, intensity and duration. Minimum value 0 maximum value 12 higher scores indicate worse craving.
Time Frame: Once per week in weeks 2 through 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 80 | 76
score on a scale | 1.12 (0.82) | 0.99 (0.71)

ADVERSE EVENTS:
Time Frame: 17 weeks
Description: Adverse events were queried at each visit.
Groups:
- Varenicline: varenicline 2 mg daily
- Placebo: Identical placebo capsules
Arm/Group | Varenicline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/76
Serious Adverse Events (participants affected / at risk) | 6/80 | 6/76
Other Adverse Events (participants affected / at risk) | 80/80 | 67/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=80) | Placebo (N=76)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lower abdominal mass (Gastrointestinal disorders) | 1 (1) | 0 (0) — Hospitalization due to lower abdominal mass
Cocaine use disorder exacerbation (Psychiatric disorders) | 1 (1) | 0 (0) — Admitted to inpatient treatment for worsening of cocaine use disorder
Substance induced depression (Psychiatric disorders) | 0 (0) | 1 (1) — Admiitted to inpatient treatment of substance induced depression
gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Admitted to inpatient treatment for gastroenteritis
orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) — admitted to inpatient treatment for orthostatic hypotension
chest pain, cocaine induced (Cardiac disorders) | 1 (1) | 0 (0) — admitted to inpatient treatment for cocaine induced chest pain
oiate detoxification (Psychiatric disorders) | 1 (1) | 0 (0) — admitted to inpatient treatment for opiate detoxification
mitral valve replacement (Cardiac disorders) | 0 (0) | 1 (1) — admitted to inpatient treatment for mitral valve replacement
chest pain (Cardiac disorders) | 1 (1) | 0 (0) — admitted to inpatient treatment for chest pain
gunshot wound (General disorders) | 0 (0) | 1 (1) — admitted to inpatient treatment for a gunshot wound
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — admitted to inpatient treatment for nausea
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=80) | Placebo (N=76)
aches and pains (Musculoskeletal and connective tissue disorders) | 20 | 23
upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 26 | 27
headache (General disorders) | 15 | 11
elevated blood pressure (Blood and lymphatic system disorders) | 14 | 11
diarrhea (Gastrointestinal disorders) | 9 | 14
abdominal pain (Gastrointestinal disorders) | 11 | 9
nausea (Gastrointestinal disorders) | 19 | 5
toothache (General disorders) | 8 | 7
vivid dreams (Nervous system disorders) | 11 | 2
fatigue (General disorders) | 5 | 7
flatulence (Gastrointestinal disorders) | 6 | 5
lightheadedness (General disorders) | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/87/NCT01680887/Prot_SAP_000.pdf